CLINICAL TRIAL: NCT06427642
Title: Efficacy Evaluation of Umbilical Cord Blood-derived Mononuclear Cells in the Treatment of Refractory Neonatal Diseases
Brief Title: Efficacy Evaluation of UCB-MNCs in the Treatment of Refractory Neonatal Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Collaborators: Qilu Children's Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNCs-2024
Record Dates: First submitted 2024-05-13; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Bronchopulmonary Dysplasia; Short Bowel Syndrome
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Bronchopulmonary Dysplasia; Short Bowel Syndrome | interventions — Parenteral Nutrition, Total

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental group for children with HIE (Experimental): Intravenous infusion of UCB-MNCs is given within 24 hours of being identified as a high-risk patient
  Interventions: Biological: Mononuclear cells; Device: Mild hypothermia therapy
- Control group for children with HIE (Active Comparator): Mild hypothermia therapy is given for 72 hours to maintain anal temperature between 33.5°C and 34°C
  Interventions: Device: Mild hypothermia therapy
- Experimental group for children with BPD (Experimental): Intravenous infusion of UCB-MNCs is given within 24 hours of being identified as a high-risk patient
  Interventions: Biological: Mononuclear cells; Device: Breathing support technique
- Control group for children with BPD (Active Comparator): Clinical routine treatment
  Interventions: Device: Breathing support technique
- Experimental group for children with SBS (Experimental): Intravenous infusion of UCB-MNCs
  Interventions: Biological: Mononuclear cells; Procedure: Total parenteral nutrition
- Control group for children with SBS (Active Comparator): Clinical routine treatment
  Interventions: Procedure: Total parenteral nutrition

INTERVENTIONS:
Biological: Mononuclear cells — UCB-MNCs are obtained from umbilical cord blood by density gradient centrifugation
  Arms: Experimental group for children with BPD; Experimental group for children with HIE; Experimental group for children with SBS
Device: Mild hypothermia therapy — Mild hypothermia therapy via hypothermia therapy apparatus
  Arms: Control group for children with HIE; Experimental group for children with HIE
Device: Breathing support technique — Breathing support via ventilator
  Arms: Control group for children with BPD; Experimental group for children with BPD
Procedure: Total parenteral nutrition — Liquid nutrition injected directly into the bloodstream
  Arms: Control group for children with SBS; Experimental group for children with SBS

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE), bronchopulmonary dysplasia (BPD), short bowel syndrome (SBS) are refractory in clinical treatment. Thus, how to better prevent such diseases is currently a key research topic in the international field. The use of cord blood-derived mononuclear cells may promote to save lives and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* For children with hypoxic-ischemic encephalopathy (HIE): meet the diagnostic criteria for HIE.

For children with bronchopulmonary dysplasia (BPD): 1) preterm infants with definite gestational age of 25-30 weeks; 2) birth weight 401-1249 g; 3) the risk of BPD was assessed to be greater than 60%. The scoring was based on the BPD high risk scoring system established by the NCHD Neonatal Cooperative Network; 4)parents read the subject's instructions, agreed to the treatment and signed the informed consent.

For children with short bowel syndrome (SBS): 1) postoperative short bowel syndrome caused by neonatal necrotizing enterocolitis and other causes (developmental malformations of the digestive tract: intestinal atresia, anal atresia, intestinal stenosis, etc.); 2) parents read the subject's instructions, agreed to the treatment and signed the informed consent.

Exclusion Criteria:

* For children with HIE: unable or unwilling to provide informed consent or unable to comply with trial requirements.

For children with BPD: 1) with severe anemia, severe intracranial hemorrhage, pulmonary hemorrhage, congenital respiratory malformations (posterior nostril atresia, tracheoesophageal fistula, cleft palate, etc.), complicated congenital heart disease, diaphragmatic hernia, shock, other serious comorbidities or complications (congenital inherited metabolic diseases, endocrine diseases, severe congenital malformations and other diseases that affect lung development); 2) unable or unwilling to provide informed consent or unable to comply with trial requirements.

For children with SBS: unable or unwilling to provide informed consent or unable to comply with trial requirements.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | Within 12 hours after UCB-MNCs infusion
  Monitor oxygen, heart rate, temperature, rash, infection, etc

SECONDARY OUTCOMES:
Incidence of complications | a year
  Children with BPD: The incidence of various complications such as pneumothorax, necrotizing enterocolitis (NEC), intraventricular hemorrhage (grade 3 and above), persistent pulmonary hypertension (PPHN), retinopathy of prematurity (ROP)
Imaging test results | 2 weeks and 6 months after UCB-MNCs infusion
  Children with HIE: Brain diffusion tensor imaging (DTI) and 18F-Fluorodeoxyglucose positron emission tomography (18F-FDG-PET/CT)
Electroencephalography (EEG) results | 7 days UCB-MNCs infusion
  Children with HIE: The frequency of seizures will be measured via EEG. Seizures appear on EEG as a sudden and transient rise in the lower and/or upper borders of amplitude
Ventilator supporting time | 1 month after UCB-MNCs infusion
  Ventilator supporting time and oxygen demand will be recorded as important indications for clinical prognosis for children with HIE or BPD
Change of Gross Motor Performance Measure (GMPM) | 1, 3, 6 months after UCB-MNCs infusion
  GMPM is a standardized measurement tool for assessing quality of movement for children with HIE. Higher value means better motor quality
Change of Gross Motor Function Measure (GMFM) | 1, 3, 6 months after UCB-MNCs infusion
  GMFM is a standardized measurement tool for assessing motor function for children with HIE. It consists of lying & rolling, sitting, crawling & kneeling, standing, etc. Higher value means better gross motor function
Biomarker of HIE | 7 days after UCB-MNCs infusion
  pNF-H, marker of central nervous system axonal damage
Biomarker of BPD | 7 days after UCB-MNCs infusion
  AGER, marker of lung epithelial cell damage
Inflammatory indicators concentrations | 7 days after UCB-MNCs infusion
  Serum IL-6, IL-8, TNF concentrations will be measured via ELISA for children with HIE, BPD or SBS

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Qilu Children's Hospital of Shandong University
Locations (1):
- Qilu Children's Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No